CLINICAL TRIAL: NCT02380222
Title: Patient-Reported Outcome Questionnaire Development for Symptoms of Systemic Mastocytosis
Brief Title: Patient-Reported Outcome Questionnaire for Systemic Mastocytosis
Status: Completed | Type: Observational
Sponsor: Adelphi Values LLC (Industry)
Collaborators: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BL7064A
Record Dates: First submitted 2015-02-26; First posted 2015-03-05 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Aggressive Systemic Mastocytosis (ASM); SM w Assoc Clonal Hema Non-mast Cell Lineage Disease (SM-AHNMD); Mast Cell Leukemia (MCL); Smoldering Systemic Mastocytosis (SSM); Indolent Systemic Mastocytosis (ISM) ISM Subgroup Fully Recruited
Keywords: Systemic mastocytosis; Patient-reported outcome (PRO)
MeSH Terms: conditions — Mastocytosis, Systemic; Leukemia, Mast-Cell | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- ASM
  Interventions: Other: Interview
- SM-AHNMD
  Interventions: Other: Interview
- MCL
  Interventions: Other: Interview
- SSM
  Interventions: Other: Interview
- ISM
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Single interview lasting approximately one hour

SUMMARY:
The purpose of this study is to explore the key symptoms of individuals with systemic mastocytosis. Interviews of enrolled individuals will be conducted to learn about the disease symptoms and condition. The interview will last approximately 60 minutes and will be conducted by a trained interviewer, be audio-recorded (with patient consent), and all information provided by the patient will be treated confidentially and made anonymous so that it is non-identifiable. The interview may be conducted face-to-face, over the phone, or virtually via Skype, a free video conferencing program, depending upon the patient's geographic location. Patients will be compensated for their participating time.

This is not a medication-related study, and no medication will be distributed or tested during this study. Participation in this study will not affect any treatment or assistance that a patient currently receives or may receive in the future.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of one of the following conditions based upon World Health Organization (WHO) diagnostic criteria: aggressive systemic mastocytosis (ASM), systemic mastocytosis with associated clonal hematologic non-mast cell lineage disease (SM-AHNMD), mast cell leukemia (MCL), smoldering systemic mastocytosis (SSM), indolent systemic mastocytosis (ISM)
* Diagnosis confirmed by bone marrow biopsy
* Fluency in English
* Willingness and ability to participate in a one-hour interview

Exclusion Criteria:

* A condition or situation that would interfere with participation in an interview (e.g., cognitive impairment or disorder, alcohol or drug abuse)
* Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness
* Any other prior malignancy except for the following: Adequately treated basal cell or squamous cell skin cancer; In situ cervical cancer; Adequately treated Stage I or II cancer from which the subject is currently in complete remission, or other cancer from which the subject has been disease-free for 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of the United States with advanced systemic mastocytosis who volunteer to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Collection of qualitative interview data on the symptoms of advanced systemic mastocytosis | Once

CONTACTS AND LOCATIONS:
Locations (1):
- Adelphi Values LLC, Boston, Massachusetts, United States